CLINICAL TRIAL: NCT02513472
Title: An Open-Label, Single-Arm Multicenter Phase 1b/2 Study to Evaluate the Efficacy and Safety of Eribulin Mesylate in Combination With Pembrolizumab in Subjects With Metastatic Triple-Negative Breast Cancer (mTNBC)
Brief Title: Study to Evaluate the Efficacy and Safety of Eribulin Mesylate in Combination With Pembrolizumab in Participants With Metastatic Triple-Negative Breast Cancer (mTNBC)
Acronym: ENHANCE-1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7389-M001-218; KEYNOTE-150 (Other: Merck Sharp and Dohme Corp)
Record Dates: First submitted 2015-07-29; First posted 2015-07-31 (Estimated); Results first posted 2020-08-14 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Breast Neoplasm
Keywords: Eribulin Mesylate; Pembrolizumab; Metastatic Triple-Negative Breast Cancer; mTNBC
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — eribulin; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Eribulin Mesylate + Pembrolizumab (Experimental): Participants with mTNBC previously treated with 0 (stratum 1) or 1 to 2 (stratum 2) lines of systemic anticancer therapy (cytotoxic or targeted anticancer agents) in the metastatic setting.
  Interventions: Drug: Eribulin Mesylate; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Eribulin Mesylate — Eribulin Mesylate will be administered as a 1.4 milligram per square meter (mg/m^2) IV (intravenous) infusion on Day 1 and Day 8 of each 21-day cycle in the presence of clinical benefit until intercurrent illness, unacceptable toxicity, or disease progression occurs, or until the participant withdraws consent.
  Other Names: Halaven, E7389
Drug: Pembrolizumab — Pembrolizumab will be administered as a 200 milligram (mg) IV infusion on Day 1 of each 21-day cycle in the presence of clinical benefit until intercurrent illness, unacceptable toxicity, or disease progression occurs, or until the participant withdraws consent.
  Other Names: Keytruda, MK-3475

SUMMARY:
This is an open-label, single-arm, multicenter, Phase 1b/2 study of eribulin mesylate in combination with pembrolizumab in participants with mTNBC previously treated with 0 (stratum 1) or 1 to 2 (stratum 2) lines of systemic anticancer therapy (cytotoxic or targeted anticancer agents) in the metastatic setting.

DETAILED DESCRIPTION:
The Phase 1b part will evaluate the safety and tolerability of eribulin mesylate in combination with pembrolizumab. Approximately 6 participants may be enrolled in the Phase 1b part of the study. The Phase 2 part will evaluate the tumor objective response rate (ORR) when treated with eribulin mesylate in combination with pembrolizumab in all participants and will also evaluate ORR in stratum 2 participants and compare with the historical response rate of pembrolizumab monotherapy 10 percent (%) in participants with mTNBC previously treated with >=1 line of prior chemotherapy in the metastatic setting. Approximately 170 mTNBC participants (including participants in Phase 1b who are on RP2D level) will be enrolled in Phase 2.

ELIGIBILITY:
Inclusion Criteria:

1. Females or males, aged >=18 years at the time of signing the informed consent form (ICF).
2. mTNBC (confirmed from most recent tissue sample) meeting the following criteria:

   1. Estrogen receptor (ER) and progesterone receptor negative (a tumor is ER and/or progesterone receptor positive if at least 1 percent (%) of the cells examined have estrogen and/or progesterone receptors) and human epidermal growth factor receptor 2 (HER2) negative (defined as immunohistochemistry [IHC] less than (<) 2+ or fluorescence in situ hybridization [FISH] negative).
   2. Previously treated with 0 to 2 lines of systemic anticancer therapy (cytotoxic or targeted anticancer agents) in the metastatic setting. Hormonal therapy and bone metastases treatment (example, bisphosphonates, denosumab, etc) are not considered forms of systemic anticancer therapy.
3. Presence of measurable disease meeting the following criteria:

   1. At least 1 lesion of >=10 millimeter (mm) in long axis diameter for nonlymph nodes or >=15 mm in short axis diameter for lymph nodes that is serially measurable according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) using computerized tomography (CT) or magnetic resonance imaging (MRI) or panoramic and close-up color photography.
   2. Lesions that have had radiotherapy must show subsequent radiographic evidence of increased size to be deemed a target lesion.
4. Life expectancy of >=3 months.
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1.
6. Adequate renal function as evidenced by serum creatinine less than or equal to (<=) 1.5 milligram per deciliter (mg/dL) or calculated creatinine clearance >=50 millimeter per minute (mL/min) according to the Cockcroft and Gault formula.
7. Adequate bone marrow function, defined as:

   1. Absolute neutrophil count (ANC) >=1.5*10^9/L.
   2. Hemoglobin (Hb) >=10.0 gram per deciliter (g/dL) (can be corrected by growth factor or transfusion).
   3. Platelet count >=100*10^9/L.
8. Adequate liver function, defined as:

   1. Total bilirubin <=1.5*upper limit of normal (ULN).
   2. Alkaline phosphatase (ALP), alanine aminotransferase (ALT), and aspartate aminotransferase (AST) <=3*ULN unless there are bone metastases, in which case liver specific alkaline phosphatase must be separated from the total and used to assess the liver function instead of the total alkaline phosphatase. ALT and AST <= 5*ULN if participant has liver metastases.
9. Resolution of all chemotherapy-related or radiation-related toxicities to Grade 1 severity or lower, except for stable sensory neuropathy (<= Grade 2) and alopecia.
10. Archived tissue sample or new biopsy sample.
11. Females must not be lactating or pregnant at Screening or Baseline (as documented by a negative beta-human chorionic gonadotropin [B-hCG] (or human chorionic gonadotropin [hCG]) test with a minimum sensitivity of 25 International units per litre (IU/L) or equivalent units of B-hCG [or hCG]). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug.
12. All females will be considered to be of childbearing potential unless they are postmenopausal (amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause) or have been sterilized surgically (that is, bilateral tubal ligation, total hysterectomy or bilateral oophorectomy, all with surgery at least 1 month before dosing).
13. Females of childbearing potential must not have had unprotected sexual intercourse within 30 days before study entry and must agree to use a highly effective method of contraception (example, total abstinence, an intrauterine device, a double-barrier method [such as condom plus diaphragm with spermicide], a contraceptive implant, a combination oral contraceptive (estrogen/progesterone), or have a vasectomized partner with confirmed azoospermia) throughout the entire study period and for 120 days after study drug discontinuation. If currently abstinent, the participant must agree to use a double barrier method as described above if she becomes sexually active during the study period or for 120 days after study drug discontinuation. Females who are using hormonal contraceptives must have been on a stable dose of the same hormonal contraceptive product for at least 28 days before dosing and must continue to use the same contraceptive during the study and for 120 days after study drug discontinuation.
14. Males who have had a successful vasectomy (confirmed azoospermia) or they and their female partners meet the criteria above (that is, not of childbearing potential or practicing highly effective contraception throughout the study period or for 120 days after study drug discontinuation). No sperm donation is allowed during the study period or for 120 days after study drug discontinuation.
15. Willing and able to comply with all aspects of the treatment protocol.
16. Provide written informed consent.

Exclusion Criteria:

1. Previous treatment with eribulin mesylate or any anti-programmed death receptor-1 (anti-PD-1), programmed death receptor ligand-1 (PD-L1), or PD-L2 agent.
2. Active autoimmune disease that has required systemic treatment in the past 2 years (that is, with use of disease modifying agents, corticosteroids, or immunosuppresive drugs). Replacement therapy (example, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc) is not considered a form of systemic treatment.
3. Less than 6 months since prior adjuvant chemotherapy.
4. Current enrollment in another interventional clinical study or used any investigational drug or device within the past 28 days preceding informed consent.
5. Treatment with chemotherapy or biological therapy within the previous 3 weeks, radiation or small molecule targeted therapy within the previous 2 weeks.
6. Known central nervous system (CNS) disease, except for those participants with treated brain metastasis who are stable for at least 1 month, having no evidence of progression or hemorrhage after treatment and no ongoing requirement for corticosteroids, as ascertained by clinical examination and brain imaging (MRI or CT) during the screening period.
7. Known history of human immunodeficiency virus (HIV) positive.
8. Known active hepatitis B (example, HBsAg reactive) or hepatitis C (example, hepatitis C virus ribonucleic acid (HCV RNA) detected).
9. Existing anticancer treatment-related toxicities of Grades >= 2 (except for alopecia and Grade 2 sensory neuropathy) according to Common Terminology Criteria for Adverse Events (CTCAE v4.03).
10. Any other malignancy that required treatment or has shown evidence of recurrence (except for nonmelanoma skin cancer, or histologically confirmed complete excision of carcinoma in situ) during the 5 years prior to enrollment in this study.
11. History of significant cardiovascular disease, defined as:

    1. congestive heart failure greater than New York Heart Association (NYHA) Class II according to the NYHA Functional Classification.
    2. unstable angina or myocardial infarction within 6 months of enrollment.
    3. serious cardiac arrhythmia.
12. Clinically significant electrocardiogram (ECG) abnormality, including a marked Baseline prolonged QT interval/corrected QT interval ([QT/QTc], example, a repeated demonstration of a QTc interval >500 millisecond [ms]).
13. History of concomitant medical conditions or infectious diseases that, in the opinion of the investigator, would compromise the participant's ability to safely complete the study.
14. Hypersensitivity to the active substance or any other excipients of the eribulin mesylate drug product, or severe hypersensitivity (>=Grade 3) to pembrolizumab and/or any of its excipients.
15. Scheduled for major surgery during the study.
16. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. The use of physiologic doses of corticosteroids may be approved after consultation with the sponsor.
17. Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
18. Has a history of interstitial lung disease.
19. Has an active infection requiring systemic therapy.
20. Has received a live-virus vaccination within 30 days of planned start of study therapy. Seasonal flu vaccines that do not contain live virus are permitted.
21. The investigator's belief that the participant is medically unfit to receive eribulin mesylate and pembrolizumab or unsuitable for any other reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2015-08-28 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2021-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Claudio Savulsky, Study Director — Eisai Inc.
Locations (22):
- United States (22):
  - Facility #1, Duarte, California
  - Facility #1, Santa Barbara, California
  - Facility #1, Denver, Colorado
  - Facility #1, Miami, Florida
  - Facility #1, West Palm Beach, Florida
  - Facility #1, Boston, Massachusetts
  - Facility #2, Boston, Massachusetts
  - Facility #1, Minneapolis, Minnesota
  - Facility #1, St Louis, Missouri
  - Facility #1, Lebanon, New Hampshire
  - Facility #1, New York, New York
  - Facility #2, New York, New York
  - Facility #1, Chattanooga, Tennessee
  - Facility #1, Nashville, Tennessee
  - Facility #1, Austin, Texas
  - Facility #1, Fort Worth, Texas
  - Facility #1, San Antonio, Texas
  - Facility #2, San Antonio, Texas
  - Facility #1, Sherman, Texas
  - Facility #1, Salem, Virginia
  - Facility #1, Winchester, Virginia
  - Facility #1, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 18 investigative sites in the United States. A total 258 participants were screened and enrolled, of which 91 were screen failures and 167 were treated. RP2D is recommended Phase 2 dose.
Pre-assignment Details: As planned, data is reported based on Stratum 1 (No prior treatment with systemic anticancer therapy) and 2 (prior 1 to 2 lines of systemic anticancer therapy) due to better estimating efficacy data for Stratum 2. All participants enrolled in Phase 1b and treated on RP2D level were pooled with the participants in Phase 2 for efficacy analysis.
Groups:
- Stratum 1: Eribulin Mesylate + Pembrolizumab: Participants with metastatic triple negative breast cancer (mTNBC) who were never treated with systemic anticancer therapy in the metastatic setting received eribulin mesylate 1.4 milligram per square meter (mg/m^2), intravenous infusion on Days 1 and 8 and pembrolizumab 200 milligram (mg), intravenous infusion on Day 1 in Treatment Cycle 1 (safety run-in, Phase 1b) and then continued in each 21-days Treatment Cycles in the presence of clinical benefit until confirmed disease progression, development of unacceptable toxicity, participant request, withdrawal of consent, or study termination by the sponsor in Phase 2 in the Stratum 1.
- Stratum 2: Eribulin Mesylate + Pembrolizumab: Participants with mTNBC previously treated with 1 to 2 lines of systemic anticancer therapy in the metastatic setting received eribulin mesylate 1.4 mg/m^2, intravenous infusion on Days 1 and 8 and pembrolizumab 200 mg, intravenous infusion on Day 1 in Treatment Cycle 1 (safety run-in, Phase 1b) and then continued in each 21-days Treatment Cycles in the presence of clinical benefit until confirmed disease progression, development of unacceptable toxicity, participant request, withdrawal of consent, or study termination by the sponsor in Phase 2 in the Stratum 2.
Period: Overall Study
Arm/Group | Stratum 1: Eribulin Mesylate + Pembrolizumab | Stratum 2: Eribulin Mesylate + Pembrolizumab
Started | 66 | 101
Phase 1b Safety run-in | 3 | 4
Phase 2 | 63 | 97
Completed | 0 | 0
Not Completed | 66 | 101
Not completed — Radiological Disease Progression | 45 | 57
Not completed — Clinical Disease Progression | 5 | 13
Not completed — Adverse Event | 8 | 11
Not completed — Withdrawal by Subject | 0 | 4
Not completed — Subject Choice | 2 | 7
Not completed — Treatment Completed as per Protocol | 3 | 3
Not completed — Other | 3 | 6

BASELINE CHARACTERISTICS:
Population: The full analysis set included all participants who received any amount of either of the study drug.
Groups:
- Stratum 1: Eribulin Mesylate + Pembrolizumab: Participants with mTNBC who were never treated with systemic anticancer therapy in the metastatic setting received eribulin mesylate 1.4 mg/m^2, intravenous infusion on Days 1 and 8 and pembrolizumab 200 mg, intravenous infusion on Day 1 in Treatment Cycle 1 (safety run-in, Phase 1b) and then continued in each 21-days Treatment Cycles in the presence of clinical benefit until confirmed disease progression, development of unacceptable toxicity, participant request, withdrawal of consent, or study termination by the sponsor in Phase 2 in the Stratum 1.
- Total: Total of all reporting groups
Arm/Group | Stratum 1: Eribulin Mesylate + Pembrolizumab | Stratum 2: Eribulin Mesylate + Pembrolizumab | Total
Number analyzed (Participants) | 66 | 101 | 167
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (10.88) | 55.6 (11.58) | 55.4 (11.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 101 | 167
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 7 | 10
  Not Hispanic or Latino | 63 | 93 | 156
  Unknown or Not Reported | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Black or African American | 7 | 12 | 19
  White | 55 | 86 | 141
  Other | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as percentage of participants with confirmed best overall response (BOR) of complete response (CR) or partial response (PR) using independent imaging review (IIR) based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. BOR of CR and PR was confirmed by a subsequent CR assessment and CR or PR assessment, respectively at least 4 weeks later. CR: disappearance of all measurable, non-measurable lesions and no unequivocal new lesions. Any pathological lymph nodes (target or non-target) had to be reduced in short axis to less than (<) 10 millimeter (mm). PR: at least a 30 percent (%) decrease in sum of diameters (SOD) of target lesions, taking as reference the baseline SOD and there are no unequivocal new lesions, and no progression of non-target disease. The 2-sided 95% confidence interval (CI) calculated by Clopper-Pearson method. As planned, data up to the primary completion date only were analyzed.
Time Frame: From date of first dose of study drug administration to date of first documentation of disease progression or death, whichever occurred first (up to 3 years 11 months)
Population: The evaluable analysis set included all participants who received any amount of either of the study drug and treated at RP2D level who had both an evaluable baseline tumor assessment and an evaluable postbaseline tumor assessment, unless discontinued early or death.
Measure: Number (95% Confidence Interval); unit: percentage of participant
Groups:
- Overall: Eribulin Mesylate + Pembrolizumab: Participants with mTNBC who were never treated with systemic anticancer therapy and previously treated with 1 to 2 lines of systemic anticancer therapy in the metastatic setting received eribulin mesylate 1.4 mg/m^2, intravenous infusion on Days 1 and 8 and pembrolizumab 200 mg, intravenous infusion on Day 1 in Treatment Cycle 1 (safety run-in, Phase 1b) and then continued in each 21-days Treatment Cycles in the presence of clinical benefit until confirmed disease progression, development of unacceptable toxicity, participant request, withdrawal of consent, or study termination by the sponsor in Phase 2 in the Stratum 1 and 2.
Arm/Group | Stratum 1: Eribulin Mesylate + Pembrolizumab | Stratum 2: Eribulin Mesylate + Pembrolizumab | Overall: Eribulin Mesylate + Pembrolizumab
Number analyzed (Participants) | 66 | 101 | 167
percentage of participant | 25.8 [15.8 to 38.0] | 21.8 [14.2 to 31.1] | 23.4 [17.2 to 30.5]

2. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was assessed by IIR based on RECIST 1.1. PFS was defined as the time from the date of the first dose of study drug to the date of the first documentation of disease progression or death, whichever occurred first. Progressive disease (PD) for target lesion, a minimum 20% increase and a minimum 5 mm absolute increase in SOD compared to nadir, or PD for non-target lesion(s) or unequivocal new lesion(s). Nadir: Lowest measure SOD of target lesion at any time point from baseline onward. The median was calculated by Kaplan-Meier (K-M) method and 95% CI were based on a generalized Brookmeyer and Crowley method. As planned, data up to the primary completion date only were analyzed.
Time Frame: as for outcome 1
Population: The full analysis set included all participants who received any amount of either of the study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stratum 1: Eribulin Mesylate + Pembrolizumab | Stratum 2: Eribulin Mesylate + Pembrolizumab | Overall: Eribulin Mesylate + Pembrolizumab
Number analyzed (Participants) | 66 | 101 | 167
months | 4.2 [3.5 to 5.5] | 4.1 [2.3 to 4.4] | 4.1 [3.5 to 4.2]

3. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of the first dose of study drug until the date of death from any cause. Median was estimated by K-M method, and the 95% CIs were based on a generalized Brookmeyer and Crowley method. As planned, data up to the primary completion date only were analyzed.
Time Frame: From date of first dose of study drug administration until date of death from any cause (up to 3 years 11 months)
Population: The full analysis set included all participants who received any amount of either of the study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stratum 1: Eribulin Mesylate + Pembrolizumab | Stratum 2: Eribulin Mesylate + Pembrolizumab | Overall: Eribulin Mesylate + Pembrolizumab
Number analyzed (Participants) | 66 | 101 | 167
months | 17.4 [13.2 to 21.0] | 15.5 [12.5 to 18.7] | 16.1 [13.3 to 18.5]

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR:time from date of confirmed OR was first documented to date of PD/death due to any cause with confirmed PR/CR using IIR as per RECIST 1.1.BOR of CR and PR was confirmed by subsequent CR assessment and CR or PR assessment, respectively at least 4 weeks later.CR:disappearance of all measurable, non-measurable lesions and no unequivocal new lesions.Any pathological lymph nodes had to be reduced in short axis to <10 mm.PR:at least 30%decrease in SOD of target lesions,taking as reference the baseline SOD, there are no unequivocal new lesions, and no progression of non-target disease.PD for target lesion, a minimum 20% increase and a minimum 5mm absolute increase in SOD compared to nadir, or PD for non-target lesions or unequivocal new lesions. Nadir:Lowest measure SOD of target lesions at any time point from baseline onward.Median calculated by K-M, 95% CI using Brookmeyer, Crowley method. As planned, data up to the primary completion date only were analyzed.
Time Frame: From the date that a confirmed objective response (OR) was first documented to the date of PD or death due to any cause for those participants with a confirmed PR or CR (up to 3 years 11 months)
Population: The full analysis set includes all participants who received any amount of either of the study drug. Here 'N' (overall number of participants analyzed) included those participants with BOR (CR or PR).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stratum 1: Eribulin Mesylate + Pembrolizumab | Stratum 2: Eribulin Mesylate + Pembrolizumab | Overall: Eribulin Mesylate + Pembrolizumab
Number analyzed (Participants) | 17 | 22 | 39
months | 9.0 [6.2 to 22.2] | 8.6 [6.2 to 25.1] | 8.3 [6.5 to 22.2]

5. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: CBR was defined as the percentage of participant, who had BOR of CR, PR, or durable stable disease (dSD) (>=24 weeks). CBR was assessed by IIR based on RECIST 1.1. BOR of CR and PR was confirmed by a subsequent CR assessment and CR or PR assessment, respectively at least 4 weeks later. CR: disappearance of all measurable, non-measurable lesions and no unequivocal new lesions. Any pathological lymph nodes (target or non-target) to be reduced in short axis to <10 mm. PR: at least a 30% decrease in SOD of target lesions, as reference the baseline SOD and no unequivocal new lesions, and no progression of non-target disease. Stable disease (SD) must be >=8 weeks after first dose date to be considered best overall response. Durable SD: subset of SD with a duration of >=24 weeks after first dose date. The 2-sided 95% CI is computed by the method of Clopper-Pearson. As planned, data up to the primary completion date only were analyzed.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participant
Arm/Group | Stratum 1: Eribulin Mesylate + Pembrolizumab | Stratum 2: Eribulin Mesylate + Pembrolizumab | Overall: Eribulin Mesylate + Pembrolizumab
Number analyzed (Participants) | 66 | 101 | 167
percentage of participant | 36.4 [24.9 to 49.1] | 29.7 [21.0 to 39.6] | 32.3 [25.3 to 40.0]

6. Secondary Outcome: ORR in the Programmed Death Receptor-Ligand 1 (PD-L1) Positive Set
Description: ORR was defined as the percentage of participant with confirmed BOR of CR or PR. ORR in the PD-L1 positive set was assessed by IIR based on RECIST 1.1. BOR of CR and PR was confirmed by a subsequent CR assessment and CR or PR assessment, respectively at least 4 weeks later. CR: disappearance of all measurable, non-measurable lesions and no unequivocal new lesions. Any pathological lymph nodes (target/non-target) to be reduced in short axis to <10 mm. PR: at least a 30% decrease in SOD of target lesions, as reference the baseline SOD and no unequivocal new lesions, and no progression of non-target disease. PD L1 status was 'Positive' if combined positive score (CPS) >=1 and 'Negative' if CPS ˂1. The 2-sided 95% CI was calculated by the method of Clopper-Pearson. As planned, data up to the primary completion date only were analyzed.
Time Frame: as for outcome 1
Population: The PD-L1 positive set included all participants who received any amount of either of the study drug, had both an evaluable baseline tumor assessment and an evaluable postbaseline tumor assessment, unless discontinued early or death and whose PD-L1 expression level was above the threshold that was to be specified prior to the final analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participant
Arm/Group | Stratum 1: Eribulin Mesylate + Pembrolizumab | Stratum 2: Eribulin Mesylate + Pembrolizumab | Overall: Eribulin Mesylate + Pembrolizumab
Number analyzed (Participants) | 29 | 45 | 74
percentage of participant | 34.5 [17.9 to 54.3] | 24.4 [12.9 to 39.5] | 28.4 [18.5 to 40.1]

7. Secondary Outcome: PFS in the PD-L1 Positive Set
Description: PFS was defined as the time from the date of the first dose of study drug to the date of the first documentation of disease progression or death, whichever occurred first. PFS in PD-L1 positive set was assessed by IIR based on RECIST 1.1. PD for target lesion, a minimum 20% increase and a minimum 5 mm absolute increase in SOD compared to nadir, or PD for non-target lesion(s) or unequivocal new lesion(s). Nadir: Lowest measure SOD of target legions at any time point from baseline onward. The median was calculated by K-M method and 95% CI are based on a generalized Brookmeyer and Crowley method. PD L1 status was 'Positive' if CPS >=1 and 'Negative' if CPS ˂1. As planned, data up to the primary completion date only were analyzed.
Time Frame: From date of first dose of study drug administration to date of first documentation of disease progression or death, whichever occurs first (up to 3 years 11 months)
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stratum 1: Eribulin Mesylate + Pembrolizumab | Stratum 2: Eribulin Mesylate + Pembrolizumab | Overall: Eribulin Mesylate + Pembrolizumab
Number analyzed (Participants) | 29 | 45 | 74
months | 6.1 [4.1 to 10.2] | 4.1 [2.1 to 4.8] | 4.2 [3.5 to 6.1]

8. Secondary Outcome: OS in the PD-L1 Positive Set
Description: OS in the PD-L1 positive set was defined as the time from the date of the first dose of study drug until the date of death from any cause. The median was estimated by KM method, and the 95% CIs were based on a generalized Brookmeyer and Crowley method. PD L1 status was 'Positive' if CPS >=1 and 'Negative' if CPS ˂1. As planned, data up to the primary completion date only were analyzed.
Time Frame: From date of first dose of study drug administration until date of death from any cause (up to 3 years 11 months)
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stratum 1: Eribulin Mesylate + Pembrolizumab | Stratum 2: Eribulin Mesylate + Pembrolizumab | Overall: Eribulin Mesylate + Pembrolizumab
Number analyzed (Participants) | 29 | 45 | 74
months | 21.0 [8.3 to 29.0] | 14.0 [11.0 to 19.4] | 16.3 [12.7 to 24.2]

9. Secondary Outcome: DOR in the PD-L1 Positive Set
Description: DOR: time from date of confirmed OR was first documented to date of PD or death due to any cause with confirmed PR or CR. DOR in PD-L1 positive set was assessed by using IIR as per RECIST 1.1. BOR of CR and PR was confirmed by a subsequent CR assessment and CR or PR assessment, respectively at least 4 weeks later. CR: disappearance of all measurable, non-measurable lesions and no unequivocal new lesions. Any pathological lymph nodes (target or non-target) had to be reduced in short axis to <10 mm. PR: at least 30%decrease in SOD of target lesions, taking as reference the baseline SOD, there are no unequivocal new lesions, and no progression of non-target disease. PD for target lesion, a minimum 20% increase and a minimum 5 mm absolute increase in SOD compared to nadir, or PD for non-target lesion(s) or unequivocal new lesion(s). Nadir: Lowest measure SOD of target lesions at any time point from baseline onward. Median calculated by K-M and 95% CI using Brookmeyer, Crowley method.
Time Frame: From the date that a confirmed objective response is first documented to the date of PD or death due to any cause for those participants with a confirmed PR or CR (up to 3 years 11 months)
Population: PD-L1 positive set:participants who received any amount of either of study drug, had both an evaluable baseline and postbaseline tumor assessment, unless discontinued early/death,whose PD-L1 expression level was above threshold that was to be specified prior to final analysis.'N'(Overall number of participants analyzed) had participants with CR/PR. As planned, data up to the primary completion date only were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stratum 1: Eribulin Mesylate + Pembrolizumab | Stratum 2: Eribulin Mesylate + Pembrolizumab | Overall: Eribulin Mesylate + Pembrolizumab
Number analyzed (Participants) | 10 | 11 | 21
months | 8.3 [3.2 to NA] — The upper limit of the 95% CI was not estimable due to the upper side of inequality is not satisfied based on Brookmeyer and Crowley method. | 8.2 [5.1 to 25.1] | 8.2 [6.2 to 25.1]

10. Other Pre Specified Outcome: CBR in the PD-L1 Positive Set
Description: CBR was defined as percentage of participant, had BOR of CR, PR, or dSD (>=24 weeks). CBR in PD-L1 positive set was assessed by IIR based on RECIST 1.1. BOR of CR and PR was confirmed by a subsequent CR assessment and CR or PR assessment, respectively at least 4 weeks later. CR: disappearance of all measurable, non-measurable lesions and no unequivocal new lesions. Any pathological lymph nodes (target or non-target) to be reduced in short axis to<10 mm. PR: at least 30 % decrease in SOD of target lesions, as reference the baseline SOD and no unequivocal new lesions, no progression of non-target disease.SD must be >=8 weeks after first dose date considered best overall response. Durable SD: subset of SD with duration of >=24 weeks after first dose date. The 2 -sided 95% CI is computed by method of Clopper-Pearson. PD L1 status was 'Positive' if CPS>=1, 'Negative' if CPS˂1. As planned, data up to the primary completion date only were analyzed.
Time Frame: as for outcome 1
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participant
Arm/Group | Stratum 1: Eribulin Mesylate + Pembrolizumab | Stratum 2: Eribulin Mesylate + Pembrolizumab | Overall: Eribulin Mesylate + Pembrolizumab
Number analyzed (Participants) | 29 | 45 | 74
percentage of participant | 48.3 [29.4 to 67.5] | 28.9 [16.4 to 44.3] | 36.5 [25.6 to 48.5]

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to 4 years 10 months
Description: Safety data is reported based on Stratums 1 and 2, and collectively for combined population participants, as planned.
Arm/Group | Stratum 1: Eribulin Mesylate + Pembrolizumab | Stratum 2: Eribulin Mesylate + Pembrolizumab | Overall: Eribulin Mesylate + Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 59/66 | 79/101 | 138/167
Serious Adverse Events (participants affected / at risk) | 30/66 | 57/101 | 87/167
Other Adverse Events (participants affected / at risk) | 66/66 | 100/101 | 166/167
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stratum 1: Eribulin Mesylate + Pembrolizumab (N=66) | Stratum 2: Eribulin Mesylate + Pembrolizumab (N=101) | Overall: Eribulin Mesylate + Pembrolizumab (N=167)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 3 | 4
Neutropenia (Blood and lymphatic system disorders) | 2 | 3 | 5
Cardiac arrest (Cardiac disorders) | 1 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 1 | 2
Retinal detachment (Eye disorders) | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 1 | 2
Constipation (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 2 | 2
Enteritis (Gastrointestinal disorders) | 0 | 1 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 3 | 3
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 1 | 2
Stomatitis (Gastrointestinal disorders) | 1 | 2 | 3
Vomiting (Gastrointestinal disorders) | 0 | 3 | 3
Asthenia (General disorders) | 0 | 3 | 3
Axillary pain (General disorders) | 0 | 1 | 1
Death (General disorders) | 1 | 1 | 2
Fatigue (General disorders) | 0 | 2 | 2
Influenza like illness (General disorders) | 0 | 1 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 2 | 4 | 6
Contrast media allergy (Immune system disorders) | 1 | 0 | 1
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 | 1 | 1
Breast cellulitis (Infections and infestations) | 0 | 2 | 2
Cellulitis (Infections and infestations) | 0 | 1 | 1
Device related infection (Infections and infestations) | 0 | 1 | 1
Herpes zoster infection neurological (Infections and infestations) | 1 | 0 | 1
Lung infection (Infections and infestations) | 0 | 1 | 1
Oesophageal candidiasis (Infections and infestations) | 1 | 1 | 2
Pneumonia (Infections and infestations) | 3 | 5 | 8
Sepsis (Infections and infestations) | 1 | 2 | 3
Septic shock (Infections and infestations) | 1 | 0 | 1
Viral myositis (Infections and infestations) | 0 | 1 | 1
Wound infection (Infections and infestations) | 0 | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 2 | 4
Wound complication (Injury, poisoning and procedural complications) | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 3 | 0 | 3
Aspartate aminotransferase increased (Investigations) | 3 | 0 | 3
Blood creatinine increased (Investigations) | 1 | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 0 | 1
Weight decreased (Investigations) | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 1 | 2
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypophagia (Metabolism and nutrition disorders) | 0 | 1 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2
Cardiac valve fibroelastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 7 | 7
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 3
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Brain oedema (Nervous system disorders) | 1 | 1 | 2
Central nervous system lesion (Nervous system disorders) | 1 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 1 | 0 | 1
Neurological symptom (Nervous system disorders) | 0 | 1 | 1
Seizure (Nervous system disorders) | 0 | 1 | 1
Subdural hygroma (Nervous system disorders) | 0 | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 2
Nephritis (Renal and urinary disorders) | 0 | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 1
Ureteric obstruction (Renal and urinary disorders) | 0 | 1 | 1
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 6
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 4
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 1
Embolism venous (Vascular disorders) | 1 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 1
Subclavian vein thrombosis (Vascular disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stratum 1: Eribulin Mesylate + Pembrolizumab (N=66) | Stratum 2: Eribulin Mesylate + Pembrolizumab (N=101) | Overall: Eribulin Mesylate + Pembrolizumab (N=167)
Anaemia (Blood and lymphatic system disorders) | 23 | 24 | 47
Neutropenia (Blood and lymphatic system disorders) | 19 | 39 | 58
Hyperthyroidism (Endocrine disorders) | 7 | 6 | 13
Hypothyroidism (Endocrine disorders) | 16 | 15 | 31
Dry eye (Eye disorders) | 2 | 7 | 9
Lacrimation increased (Eye disorders) | 6 | 8 | 14
Vision blurred (Eye disorders) | 4 | 7 | 11
Abdominal distension (Gastrointestinal disorders) | 4 | 8 | 12
Abdominal pain (Gastrointestinal disorders) | 9 | 15 | 24
Abdominal pain upper (Gastrointestinal disorders) | 5 | 7 | 12
Constipation (Gastrointestinal disorders) | 29 | 33 | 62
Diarrhoea (Gastrointestinal disorders) | 19 | 33 | 52
Dry mouth (Gastrointestinal disorders) | 11 | 16 | 27
Dyspepsia (Gastrointestinal disorders) | 11 | 9 | 20
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 6 | 11
Nausea (Gastrointestinal disorders) | 45 | 51 | 96
Stomatitis (Gastrointestinal disorders) | 7 | 25 | 32
Vomiting (Gastrointestinal disorders) | 18 | 26 | 44
Asthenia (General disorders) | 5 | 7 | 12
Chills (General disorders) | 9 | 9 | 18
Fatigue (General disorders) | 48 | 63 | 111
Influenza like illness (General disorders) | 4 | 6 | 10
Non-cardiac chest pain (General disorders) | 1 | 8 | 9
Oedema peripheral (General disorders) | 8 | 7 | 15
Pyrexia (General disorders) | 22 | 29 | 51
Upper respiratory tract infection (Infections and infestations) | 8 | 9 | 17
Urinary tract infection (Infections and infestations) | 10 | 19 | 29
Fall (Injury, poisoning and procedural complications) | 3 | 8 | 11
Alanine aminotransferase increased (Investigations) | 15 | 11 | 26
Aspartate aminotransferase increased (Investigations) | 15 | 14 | 29
Blood alkaline phosphatase increased (Investigations) | 3 | 9 | 12
Blood creatinine increased (Investigations) | 3 | 7 | 10
Neutrophil count decreased (Investigations) | 10 | 12 | 22
Platelet count decreased (Investigations) | 4 | 5 | 9
Weight decreased (Investigations) | 20 | 21 | 41
White blood cell count decreased (Investigations) | 6 | 13 | 19
Decreased appetite (Metabolism and nutrition disorders) | 29 | 23 | 52
Dehydration (Metabolism and nutrition disorders) | 11 | 16 | 27
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 8 | 11
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 9 | 10
Hypokalaemia (Metabolism and nutrition disorders) | 15 | 13 | 28
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 | 13 | 18
Hyponatraemia (Metabolism and nutrition disorders) | 6 | 13 | 19
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 | 22 | 46
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 20 | 26
Bone pain (Musculoskeletal and connective tissue disorders) | 5 | 4 | 9
Flank pain (Musculoskeletal and connective tissue disorders) | 3 | 6 | 9
Muscle spasms (Musculoskeletal and connective tissue disorders) | 10 | 6 | 16
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 | 5 | 10
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 12 | 7 | 19
Myalgia (Musculoskeletal and connective tissue disorders) | 11 | 9 | 20
Neck pain (Musculoskeletal and connective tissue disorders) | 7 | 4 | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 | 14 | 24
Dizziness (Nervous system disorders) | 13 | 15 | 28
Dysgeusia (Nervous system disorders) | 6 | 8 | 14
Headache (Nervous system disorders) | 22 | 20 | 42
Hypoaesthesia (Nervous system disorders) | 7 | 3 | 10
Paraesthesia (Nervous system disorders) | 4 | 5 | 9
Peripheral sensory neuropathy (Nervous system disorders) | 35 | 34 | 69
Taste disorder (Nervous system disorders) | 6 | 3 | 9
Anxiety (Psychiatric disorders) | 6 | 7 | 13
Depression (Psychiatric disorders) | 6 | 7 | 13
Insomnia (Psychiatric disorders) | 11 | 11 | 22
Breast pain (Reproductive system and breast disorders) | 4 | 3 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 24 | 31 | 55
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 | 23 | 39
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 9 | 9 | 18
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 7 | 14
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 9 | 13
Alopecia (Skin and subcutaneous tissue disorders) | 35 | 31 | 66
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 12 | 21
Rash (Skin and subcutaneous tissue disorders) | 16 | 14 | 30
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9 | 9 | 18
Hot flush (Vascular disorders) | 10 | 11 | 21
Hypertension (Vascular disorders) | 3 | 9 | 12
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 7 | 7
Oral candidiasis (Infections and infestations) | 4 | 3 | 7
Sinusitis (Infections and infestations) | 2 | 6 | 8
Arthritis (Musculoskeletal and connective tissue disorders) | 5 | 1 | 5
Joint swelling (Musculoskeletal and connective tissue disorders) | 5 | 1 | 6
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 | 5 | 9
Memory impairment (Nervous system disorders) | 4 | 2 | 6
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 7
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 0 | 4
Hypotension (Vascular disorders) | 4 | 4 | 8
Leukopenia (Blood and lymphatic system disorders) | 4 | 4 | 8
Blood bilirubin increased (Investigations) | 4 | 1 | 5
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-26): https://cdn.clinicaltrials.gov/large-docs/72/NCT02513472/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-08): https://cdn.clinicaltrials.gov/large-docs/72/NCT02513472/SAP_001.pdf